CLINICAL TRIAL: NCT04827732
Title: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) in the Reirradiation of Locoregionally Recurrent Rectal Cancer - IMPARC
Brief Title: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) in Recurrent Rectal Cancer
Acronym: IMPARC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202103218
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (Experimental): * Radiotherapy will consist of five fractions, delivered once daily, with pencil beam scanning proton beam therapy using the defined dose in dose level 1 (30 Gy).
  * The use of Intensity Modulated Radiation Therapy (IMRT) with photon beam therapy is permitted at the discretion of the treating investigator in order to avoid extended treatment delays due to logistical reasons (e.g. machine downtime).
  Interventions: Radiation: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy; Device: MEVION S250i Hyperscan and Adaptive Aperture Proton Therapy Machine
- Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (Experimental): * Radiotherapy will consist of five fractions, delivered once daily, with pencil beam scanning proton beam therapy using the defined dose in dose level 2 (35 Gy).
  * The use of Intensity Modulated Radiation Therapy (IMRT) with photon beam therapy is permitted at the discretion of the treating investigator in order to avoid extended treatment delays due to logistical reasons (e.g. machine downtime).
  Interventions: Radiation: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy; Device: MEVION S250i Hyperscan and Adaptive Aperture Proton Therapy Machine
- Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (Experimental): * Radiotherapy will consist of five fractions, delivered once daily, with pencil beam scanning proton beam therapy using the defined dose in dose level 3 (40 Gy).
  * The use of Intensity Modulated Radiation Therapy (IMRT) with photon beam therapy is permitted at the discretion of the treating investigator in order to avoid extended treatment delays due to logistical reasons (e.g. machine downtime).
  Interventions: Radiation: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy; Device: MEVION S250i Hyperscan and Adaptive Aperture Proton Therapy Machine
- Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (Experimental): * Radiotherapy will consist of five fractions, delivered once daily, with pencil beam scanning proton beam therapy using the defined dose in dose level -1 (25 Gy).
  * The use of Intensity Modulated Radiation Therapy (IMRT) with photon beam therapy is permitted at the discretion of the treating investigator in order to avoid extended treatment delays due to logistical reasons (e.g. machine downtime).
  Interventions: Radiation: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy; Device: MEVION S250i Hyperscan and Adaptive Aperture Proton Therapy Machine

INTERVENTIONS:
Radiation: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy — When feasible it is strongly recommended that radiotherapy begin on a Monday
  Other Names: IMPT
Device: MEVION S250i Hyperscan and Adaptive Aperture Proton Therapy Machine — -The device that will administer the IMPT

SUMMARY:
The purpose of this trial is to determine the maximum tolerated dose (MTD) of hypofractionated IMPT for the reirradiation of locoregionally recurrent rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* History of biopsy-proven adenocarcinoma of the rectum, anus or rectosigmoid junction of any stage now with recurrent disease in the pelvis
* One prior course of radiation therapy to the pelvis for rectal cancer
* ECOG performance status 0-2
* At least 18 years of age
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Patients with pre-existing radiosensitizing conditions, such as connective tissue disorders (i.e. lupus, scleroderma) and genetic mutations (i.e. ataxia-telangiectasia)
* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease, basal cell or squamous cell carcinoma of the skin that were treated with local resection only, or carcinoma in situ of the cervix. Patients with history of prostate cancer treated without radiotherapy and no evidence of disease are eligible
* More than one prior course of radiation to the pelvis for rectal cancer
* Prior radiation to the pelvis for disease other than rectal cancer
* Tumor in the rectum/colon requiring radiation therapy to the full circumference of the rectum/colon.
* Current treatment with any investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or unstable angina pectoris
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative urine or serum pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Waters, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Started | 1 | 7 | 3 | 4
Completed | 1 | 6 | 3 | 3
Not Completed | 0 | 1 | 0 | 1
Not completed — Did not start treatment | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Total
Number analyzed (Participants) | 7 | 3 | 4 | 1 | 15
Age, Continuous [Median (Full Range); unit: years] | 55 [43 to 79] | 66 [27 to 68] | 67 [49 to 69] | 54 [54 to 54] | 56 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 0 | 5
  Male | 6 | 2 | 1 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 3 | 3 | 1 | 14
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 3 | 4 | 1 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 4 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Reirradiation Using Hypofractionated IMPT
Description: * MTD is defined as the dose associated with a 35% probability of dose-limiting toxicity (DLT).
  * DLT is defined as any toxicity listed below that occurs within 6 months from start of treatment and is considered possibly, probably, or definitely related to proton reirradiation:
    * Any grade 5 toxicities
    * Any grade 4-5 GI toxicities
    * Bowel obstruction
    * Grade 3-5: diarrhea; anal, colonic, or bowel ulcers; bladder perforation; any fistula formations; peripheral motor/sensory neuropathy of the pelvis above baseline; osteonecrosis/soft tissue necrosis; radiation dermatitis; hematuria; hematochezia; bowel/pelvic hemorrhage; reproductive tract toxicity
  * Toxicity will be graded using CTCAE v5
Time Frame: From start of treatment through 6 months
Population: 3 participants are not evaluable for this outcome measure. 2 participants did not start treatment. 1 participant was erroneously treated with dose level -1 (25 Gy) which is not part of the dose levels defined in the protocol.
Measure: Number; unit: GY in 5 fractions
Groups:
- All Dose Levels: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT): * Radiotherapy will consist of five fractions, delivered once daily, with pencil beam scanning proton beam therapy using the defined dose in dose level 1 (30 Gy), dose level 2 (35 Gy), and dose level 3 (40 Gy).
  * The use of Intensity Modulated Radiation Therapy (IMRT) with photon beam therapy is permitted at the discretion of the treating investigator in order to avoid extended treatment delays due to logistical reasons (e.g. machine downtime).
Arm/Group | All Dose Levels: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 12
GY in 5 fractions | 40

2. Secondary Outcome: Clinical Complete Response Rate
Description: -DRE, endoscopy, and cross-sectional imaging will be used to measure clinical complete response rate
Time Frame: Within 6 weeks to 3 months post-completion of radiation therapy (range 7-14 weeks)
Population: 1 participant is not evaluable in Dose Level 1 because they did not start treatment. 1 participant is not evaluable in Dose Level 3 because they did not start treatment. 1 participant was erroneously treated with dose level -1 (25 Gy) which is not part of the dose levels defined in the protocol and was excluded from this outcome measure as data was not collected on the patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 6 | 3 | 3 | 0
Participants | 0 | 0 | 0 |

3. Secondary Outcome: Median Freedom From Locoregional Progression (FFLP)
Description: -Defined as time from end of radiation therapy to date of first instance of local or regional tumor progression
Time Frame: Through completion of follow-up (full range 1.81 months-13.87 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 6 | 3 | 3 | 0
months | 7.53 [1.81 to 13.87] | 9.53 [2.01 to 10.72] | 4.37 [4.01 to 12.72] |

4. Secondary Outcome: Median Overall Survival (OS)
Description: Defined as time from end of radiation therapy to date that at least 50% of patients died
Time Frame: Through completion of follow-up (full range 4.4 months to 13.87 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 6 | 3 | 3 | 0
months | NA [6.4 to 13.87] — Median overall survival not reached as at least 50% of the participants are still alive | 9.53 [8.58 to 10.72] | NA [4.4 to 12.72] — Median overall survival not reached as at least 50% of the participants are still alive |

5. Secondary Outcome: Median Progression-free Survival (PFS)
Description: -Defined as time from end of radiation therapy to the earliest date of locoregional progression, distant progression, or death from any cause
Time Frame: Through completion of follow-up (full range 1.81 months-13.87 months)
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 6 | 3 | 3 | 0
months | 2.04 [1.32 to 13.87] | 9.53 [2.01 to 10.72] | 4.37 [4.01 to 12.72] |

6. Secondary Outcome: Median Change in Quality of Life (QoL) Score as Measured by The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: 30 question survey which assesses patient well-being with 5 functional scales, 9 symptom scales, & global health scale. Scores for each scale range from 0-100. Higher score for the functional scale & global health represent high functioning, while high score for symptom scale represents high symptomatology. Median scores were taken for each scale for each dose level and the different between pre-treatment and post-treatment scores were calculated to determine change in score over time. For functional scales and global health status, negative values represent improved functionality/quality of life, while positive values represent diminished functionality. For symptom scales, the opposite is true. If patients did not complete the the survey at each time point, their data was censored. Data values were averaged prior to 3 months. Differences were taken between baseline values and the average value calculated of post-RT up to 3 months.
Time Frame: Assessed at pre-treatment (baseline), 1-2 weeks, 3 months, 6 months, 9 months, and 12 months post-treatment
Population: This outcome measure includes data for participants who completed the questionnaire. If a participant did not complete the questionnaire at a specific time point, then the participant is not included in the number analyzed at that time point. 1 participant was erroneously treated with dose level -1 (25 Gy) which is not part of the dose levels defined in the protocol and was excluded from this outcome measure as data was not collected on the participant.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 4 | 3 | 1 | 0
score on a scale
  Global health status | -4.17 [-25 to 16.67] | 0 [-33.3 to 16.67] | 8.34 [8.34 to 8.34] |
  Physical functioning | 0 [0 to 0] | 6.67 [0 to 13.33] | -6.67 [-6.67 to -6.67] |
  Role functioning | 0 [0 to 0] | 0 [0 to 0] | -16.67 [-16.67 to -16.67] |
  Emotional functioning | -6.67 [-20 to 0] | 0 [-33.33 to 6.67] | 6.67 [6.67 to 6.67] |
  Cognitive functioning | -8.33 [-16.67 to 0] | 0 [-33.3 to 16.67] | -16.67 [-16.67 to -16.67] |
  Social functioning | 8.33 [0 to 50] | 0 [0 to 0] | -33.33 [-33.33 to -33.33] |
  Fatigue | 0 [-22.2 to 0] | 0 [-11.11 to 22.22] | 0 [0 to 0] |
  Nausea and vomiting | 0 [0 to 0] | 0 [-16.67 to 0] | 16.67 [16.67 to 16.67] |
  Pain | 0 [0 to 0] | -16.67 [-16.67 to 33.33] | 16.66 [16.66 to 16.66] |
  Dyspnea | 0 [-33.3 to 0] | 0 [0 to 0] | 33.33 [33.33 to 33.33] |
  Insomnia | 0 [-33.33 to 33.33] | 0 [0 to 0] | 0 [0 to 0] |
  Appetite loss | 0 [0 to 33.33] | 0 [0 to 0] | 33.33 [33.33 to 33.33] |
  Constipation | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] |
  Diarrhea | 16.67 [0 to 33.33] | 0 [-33.33 to 33.33] | 33.33 [33.33 to 33.33] |
  Financial difficulties | 0 [0 to 66.67] | 0 [-33.33 to 0] | 33.33 [33.33 to 33.33] |

7. Secondary Outcome: Median Change in Quality of Life (QoL) Score as Measured by The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30)
Description: 30 question survey which assesses patient well-being with 5 functional scales, 9 symptom scales, & global health scale. Scores for each scale range from 0-100. Higher score for the functional scale & global health represent high functioning, while high score for symptom scale represents high symptomatology. Median scores were taken for each scale for each dose level and the different between pre-treatment and post-treatment scores were calculated to determine change in score over time. For functional scales and global health status, negative values represent improved functionality/quality of life, while positive values represent diminished functionality. For symptom scales, the opposite is true. If patients did not complete the survey at each time point, their data was censored. Data values were averaged from 3-12 months. Differences were taken between baseline values and the average value calculated of post-RT from 3-12 months.
Time Frame: Assessed at pre-treatment (baseline), 1-2 weeks, 3 months, 6 months, 9 months, and 12 months post-treatment
Population: as for outcome 6
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 4 | 3 | 1 | 0
score on a scale
  Global health status | 8.33 [0 to 54.17] | 0 [-22.22 to 0] | 8.33 [8.33 to 8.33] |
  Physical functioning | 3.33 [0 to 26.67] | 2.22 [0 to 3.33] | 0 [0 to 0] |
  Role functioning | 16.67 [0 to 58.33] | 11.11 [0 to 33.33] | 0 [0 to 0] |
  Emotional functioning | -3.33 [-16.67 to 20] | -2.22 [-10 to 0] | -10 [-10 to -10] |
  Cognitive functioning | 0 [-16.67 to 8.33] | -8.33 [-16.67 to 0] | -8.34 [-8.34 to -8.34] |
  Social functioning | 8.33 [0 to 16.67] | 5.56 [0 to 16.67] | -25 [-25 to -25] |
  Fatigue | -19.44 [-61.11 to -5.56] | 5.56 [0 to 25.93] | 0 [0 to 0] |
  Nausea and vomiting | 0 [-8.33 to 0] | 0 [-5.56 to 8.33] | -8.33 [-8.33 to -8.33] |
  Pain | -10.42 [-75 to 0] | 25 [-33.33 to 27.78] | 16.66 [16.66 to 16.66] |
  Dyspnea | -16.67 [-100 to 0] | 0 [-16.67 to 33.33] | 16.66 [16.66 to 16.66] |
  Insomnia | -25 [-33.33 to -8.33] | 0 [-11.11 to 16.67] | 33.34 [33.34 to 33.34] |
  Appetite loss | 0 [0 to 0] | 0 [-33.33 to 0] | 0 [0 to 0] |
  Constipation | -16.67 [-33.33 to 0] | 0 [-11.11 to 0] | -16.67 [-16.67 to -16.67] |
  Diarrhea | 0 [-16.67 to 0] | 0 [-50 to 33.33] | 0 [0 to 0] |
  Financial difficulties | 0 [-33.33 to 66.67] | 0 [0 to 33.33] | 16.67 [16.67 to 16.67] |

8. Secondary Outcome: Median Change in Quality of Life (QoL) Score as Measured by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer Module 29 (EORTC QLQ-CR29)
Description: 29 question survey which assesses quality of life for patients with colorectal cancer including functional & symptom status. The survey includes 4 multi-item scales & 19 single-item scales. Scores are linearly transformed to provide a score from 0-100. A high score for functional scales represents high level of functioning, while a high score for symptom scale represents high level of symptoms. Median scores were taken for each scale & the difference between baseline & varying time points was reported. Negative value represents improved function for a functional scale item, & worsening symptoms for symptom scale items. Positive values represent the converse. If patients did not complete the survey at each time point, their data was censored. Data values were averaged prior to 3 months. Differences were taken between pre-treatment (baseline) values and the average value calculated of post-RT up to 3 months.
Time Frame: Assessed at pre-treatment (baseline), 1-2 weeks, 3 months, 6 months, 9 months, and 12 months post-treatment
Population: as for outcome 6
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 4 | 3 | 1 | 0
score on a scale
  Anxiety | 0 [-33.33 to 33.33] | 0 [0 to 0] | -33.34 [-33.34 to -33.34] |
  Body image | -12.5 [-25 to 0] | 8.33 [-16.67 to 8.33] | 8.34 [8.34 to 8.34] |
  Male sexual function: number analyzed (Participants) | 3 | 2 | 0 | 0
  Male sexual function | 0 [-66.67 to 66.67] | -16.67 [-33.33 to 0] |  |
  Female sexual function: number analyzed (Participants) | 1 | 1 | 1 | 0
  Female sexual function | 0 [0 to 0] | 0 [0 to 0] | -33.33 [-33.33 to -33.33] |
  Micturition | 4.17 [-8.33 to 8.33] | -8.33 [-25 to 0] | 8.33 [8.33 to 8.33] |
  Abdominal and pelvic pain | 0 [0 to 16.67] | -16.67 [-33.33 to 33.33] | 0 [0 to 0] |
  Bloated feeling | 0 [0 to 0] | 0 [0 to -3.33] | 0 [0 to 0] |
  Dry mouth | 0 [0 to 3.33] | 0 [-33.33 to 33.33] | -33.34 [-33.34 to -33.34] |
  Hair loss | 0 [0 to 66.67] | 0 [0 to 0] | -66.67 [-66.67 to -66.67] |
  Trouble with taste | 0 [0 to 0] | -33.3 [-66.6 to 0] | 33.34 [33.34 to 33.34] |
  Stoma related problems: number analyzed (Participants) | 3 | 2 | 1 | 0
  Stoma related problems | 11.11 [0 to 16.67] | 0 [0 to 0] | 5.56 [5.56 to 5.56] |
  Defecation problems | 0 [0 to 16.67] | 0 [-16.67 to 0] | 0 [0 to 0] |
  Fecal incontinence: number analyzed (Participants) | 1 | 0 | 0 | 0
  Fecal incontinence | 16.67 [16.67 to 16.67] |  |  |
  Sore skin: number analyzed (Participants) | 1 | 0 | 0 | 0
  Sore skin | 0 [0 to 0] |  |  |
  Embarrassed by bowel movements: number analyzed (Participants) | 1 | 0 | 0 | 0
  Embarrassed by bowel movements | 33.34 [33.34 to 33.34] |  |  |
  Impotence: number analyzed (Participants) | 3 | 1 | 0 | 0
  Impotence | 0 [0 to 0] | 0 [0 to 0] |  |
  Dyspareunia: number analyzed (Participants) | 1 | 0 | 1 | 0
  Dyspareunia | -33.33 [-33.33 to -33.33] |  | 0 [0 to 0] |

9. Secondary Outcome: Median Change in Quality of Life (QoL) Score as Measured by the by the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer Module 29 (EORTC QLQ-CR29)
Description: 29 question survey which assesses quality of life for patients with colorectal cancer including functional & symptom status. The survey includes 4 multi-item scales & 19 single-item scales. Scores are linearly transformed to provide a score from 0-100. A high score for functional scales represents high level of functioning, while a high score for symptom scale represents high level of symptoms. Median scores were taken for each scale & the difference between baseline & varying time points was reported. Negative value represents improved function for a functional scale item, & worsening symptoms for symptom scale items. Positive values represent the converse. If patients did not complete the survey at each time point, their data was censored. Data values were averaged from 3-12 months. Differences were taken between baseline values and the average value calculated of post-RT from 3-12 months
Time Frame: Assessed at pre-treatment (baseline), 1-2 weeks, 3 months, 6 months, 9 months, and 12 months post-treatment
Population: as for outcome 6
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 4 | 3 | 1 | 0
score on a scale
  Anxiety | 8.33 [-8.33 to 16.67] | 0 [0 to 0] | -16.67 [-16.67 to -16.67] |
  Body image | 1.04 [-16.67 to 20.83] | -8.33 [-22.22 to 8.33] | 4.17 [4.17 to 4.17] |
  Male sexual function: number analyzed (Participants) | 3 | 2 | 0 | 0
  Male sexual function | 0 [0 to 0] | -16.67 [-33.33 to 0] |  |
  Female sexual function: number analyzed (Participants) | 1 | 1 | 1 | 0
  Female sexual function | 8.34 [8.34 to 8.34] | 0 [0 to 0] | -33.33 [-33.33 to -33.33] |
  Micturition | 0 [-12.5 to 8.33] | -19.44 [-41.67 to 16.67] | 4.16 [4.16 to 4.16] |
  Abdominal and pelvic pain | -8.33 [-75 to 0] | 0 [0 to 22.22] | -8.33 [-8.33 to -8.33] |
  Bloated feeling | 0 [-33.33 to 0] | 0 [-33.33 to 0] | 0 [0 to 0] |
  Dry mouth | 0 [-33.33 to 33.33] | 0 [-16.67 to 0] | 16.66 [16.66 to 16.66] |
  Hair loss | 0 [-33.33 to 66.67] | 0 [-77.78 to 16.67] | -33.33 [-33.33 to -33.33] |
  Trouble with taste | 0 [0 to 0] | -33.33 [-50 to -22.22] | 50 [50 to 50] |
  Stoma related problems: number analyzed (Participants) | 3 | 2 | 1 | 0
  Stoma related problems | 2.78 [-8.33 to 13.89] | -5.56 [-11.11 to 0] | 5.56 [5.56 to 5.56] |
  Defecation problems | 0 [0 to 8.33] | 0 [-22.22 to 0] | 0 [0 to 0] |
  Fecal incontinence: number analyzed (Participants) | 1 | 0 | 0 | 0
  Fecal incontinence | 16.67 [16.67 to 16.67] |  |  |
  Sore skin: number analyzed (Participants) | 1 | 0 | 0 | 0
  Sore skin | 0 [0 to 0] |  |  |
  Embarrassed by bowel movements: number analyzed (Participants) | 1 | 0 | 0 | 0
  Embarrassed by bowel movements | 33.34 [33.34 to 33.34] |  |  |
  Impotence: number analyzed (Participants) | 3 | 1 | 0 | 0
  Impotence | 0 [0 to 0] | -33.3 [-33.3 to -33.3] |  |
  Dyspareunia: number analyzed (Participants) | 1 | 0 | 1 | 0
  Dyspareunia | -33.34 [-33.34 to -33.34] |  | 0 [0 to 0] |

10. Secondary Outcome: Frequency of Treatment-related Acute Adverse Events as Measured by CTCAE v 5.0
Time Frame: From start of treatment through 3 months after completion of radiation therapy (estimated to be 3 months and 1 week)
Population: 1 participant is not evaluable in Dose Level 1 because they did not start treatment. 1 participant is not evaluable in Dose Level 3 because they did not start treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 6 | 3 | 3 | 1
Participants
  Fatigue | 1 | 1 | 2 | 0
  Dyspareunia | 1 | 0 | 0 | 0
  Pelvic pressure | 0 | 1 | 0 | 0
  Vaginal dryness | 1 | 0 | 0 | 0
  Erectile dysfunction | 1 | 0 | 0 | 0
  Scrotal pain | 0 | 1 | 0 | 0
  Urinary urgency | 2 | 0 | 0 | 0
  Urinary retention | 1 | 0 | 0 | 0
  Bladder spasm | 1 | 0 | 0 | 0
  Dysuria | 1 | 0 | 0 | 0
  Diarrhea | 1 | 1 | 1 | 1
  Dehydration | 0 | 1 | 0 | 0
  Nausea | 0 | 1 | 0 | 0
  Constipation | 0 | 1 | 0 | 0
  Small intestinal obstruction | 0 | 1 | 0 | 0
  Rectal bleeding | 0 | 0 | 1 | 0
  Buttock pain | 0 | 1 | 0 | 0

11. Secondary Outcome: Frequency of Treatment-related Late Adverse Events as Measured by CTCAE v 5.0
Time Frame: From 3 month post-completion of radiation therapy to 12 months post-completion of radiation therapy
Population: 1 participant is not evaluable in Dose Level 1 because they did not start treatment. 1 participant is not evaluable in Dose Level 3 because they did not start treatment. 1 participants in Dose Level -1 is not evaluable as patient did not have follow-up to evaluate for late adverse effects.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
Number analyzed (Participants) | 6 | 3 | 3 | 0
Participants
  Anemia | 1 | 0 | 0 |
  Fatigue | 1 | 0 | 1 |
  Urinary tract obstruction | 0 | 1 | 0 |
  Urinary incontinence | 0 | 1 | 0 |
  Nausea | 1 | 0 | 0 |
  Abdominal pain | 1 | 0 | 1 |
  Constipation | 1 | 0 | 0 |
  Rectal pain | 1 | 0 | 0 |
  Rectal perforation | 1 | 0 | 0 |
  Ischemic bowel | 1 | 0 | 0 |
  Rectal stump dehiscence | 1 | 0 | 0 |
  Stool leakage | 1 | 1 | 0 |
  Small intestinal obstruction | 1 | 0 | 1 |
  Diarrhea | 0 | 0 | 1 |
  Anorexia | 1 | 1 | 0 |
  Myalgia | 0 | 0 | 0 |
  Back pain | 0 | 0 | 1 |
  Pain in extremity | 0 | 0 | 1 |
  Generalized weakness | 0 | 0 | 1 |
  Muscle ache | 0 | 0 | 1 |
  Peripheral neuropathy | 0 | 0 | 1 |
  Fall | 0 | 0 | 1 |
  Ulceration (ankle) | 0 | 0 | 1 |
  Alopecia | 1 | 0 | 0 |
  Leaking abscess | 0 | 1 | 0 |
  Lymphedema | 0 | 0 | 1 |

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected through completion of follow-up (full range 4.4 months through 13.87 months). Adverse events were collected from start of treatment through 12 months after completion of radiation therapy.
Arm/Group | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT)
All-Cause Mortality (participants affected / at risk) | 0/1 | 2/6 | 2/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 4/6 | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 1/1 | 6/6 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=1) | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=6) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=3) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ischemic bowel (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Redness and drainage around buttocks wound (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Chronic abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Pelvic abscess (complication from surgery) (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Death due to disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level -1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=1) | Dose Level 1: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=6) | Dose Level 2: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=3) | Dose Level 3: Hypofractionated Pencil-Beam Scanning Intensity-modulated Proton Therapy (IMPT) (N=3)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Scleral disorder (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Full feeling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth sore (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 2
Rectal bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rectal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal frequency and urgency (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Stool leakage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Cold sensitivity (General disorders) | 0 | 0 | 0 | 2
Fatigue (General disorders) | 1 | 2 | 2 | 2
Fever (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 5 | 0 | 0
COVID-19 infection (Infections and infestations) | 0 | 1 | 0 | 0
Mass or abscess with leaking (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood lactacte dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Muscle ache/tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Sciatic pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumor reopened after radiation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral motor neutropathy (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urinary hesitancy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 3 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Pelvic pressure (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Skin tingling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT04827732/Prot_SAP_002.pdf